CLINICAL TRIAL: NCT01143844
Title: Assessing Fertility Potential in Female Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 804237; UPCC12807 (Other: University of Pennsylvania Abramson Cancer Center)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Effects of Chemotherapy
Keywords: Oncofertility; Fertility; Late effects; cancer; chemotherapy; radiation therapy; survivor; ovarian reserve; premature ovarian failure; early menopause; healthy volunteers; perimenopause; middle age; pediatric survivors; healthy women
MeSH Terms: conditions — Neoplasms; Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exposed females, ages 11-40: * Prior exposure to alkylating agent chemotherapy and/or radiation therapy
  * At least 1 year from completion of chemotherapy and/or radiation therapy
  * Uterus and at least one ovary are present
  * Not pregnant or breastfeeding in the past 3 months
  * Not taking any hormones or oral contraceptives for at least 4 weeks prior to study visits
  * No medical condition (other than cancer) known to be associated with premature ovarian failure (such as Turner's Syndrome or Fragile X) or ovulatory dysfunction (such as thyroid disease, congenital adrenal hyperplasia, Cushing's syndrome, hyperprolactinemia, and polycystic ovary syndrome).
- Unexposed females, ages 40-50: * Never exposed to chemotherapy or radiation therapy
  * Regular menstrual cycle (every 21-35 days)
  * Uterus and at least one ovary are present
  * Not pregnant or breastfeeding in the past 3 months
  * Not taking any hormones or oral contraceptives for at least 4 weeks prior to study visits
  * No medical condition known to be associated with premature ovarian failure (such as Turner's Syndrome or Fragile X) or ovulatory dysfunction (such as thyroid disease, congenital adrenal hyperplasia, Cushing's syndrome, hyperprolactinemia, and polycystic ovary syndrome).
- Unexposed females, ages 11-35: * Never exposed to chemotherapy or radiation therapy
  * Regular menstrual cycle (every 21-35 days)
  * Uterus and at least one ovary are present
  * Not pregnant or breastfeeding in the past 3 months
  * Not taking any hormones or oral contraceptives for at least 4 weeks prior to study visits
  * No medical condition known to be associated with premature ovarian failure (such as Turner's Syndrome or Fragile X) or ovulatory dysfunction (such as thyroid disease, congenital adrenal hyperplasia, Cushing's syndrome, hyperprolactinemia, and polycystic ovary syndrome).

SUMMARY:
Hypothesis: Girls and women exposed to chemotherapy and/or radiation therapy experience endocrine changes more similar to women in their late reproductive years than to same-age peers. These changes will be more dramatic in women who receive high dose therapy compared to women who receive low dose therapy.

At annual visits over 3-5 years, a combination of physical exam, medical history, menstrual diary keeping, pelvic ultrasound and blood hormones tests will be used to measure "ovarian reserve" , that is the number and quality of the eggs that remain in the ovaries. The study will also try to learn if those who received higher doses of certain chemotherapies are more likely to have changes in these tests sooner than those women who received smaller doses of these same drugs. Additionally a DNA (deoxyribonucleic acid) sample will be collected to look for gene variations that may predict susceptibility to ovarian damage from cancer treatments. Information learned from this study may help researchers to develop guidelines to identify problems with a female cancer survivor's ovaries before irregular menses or other symptoms of ovarian failure occur.

DETAILED DESCRIPTION:
Up to 400 females will participate in this study in one of three cohorts:

* 150 females ages 11-35, with history of exposure to alkylating agent chemotherapy and/or radiation therapy
* 150 Unexposed peers, ages 11-35, never exposed to chemotherapy or radiation therapy
* 100 Unexposed females, ages 40-50 never exposed to chemotherapy or radiation therapy

ELIGIBILITY:
Inclusion Criteria for cancer survivors:

* Previous treatment with chemotherapy and/or radiation therapy for either cancer or another illness.
* Age between 11-35 years.
* Post-menarchal.
* Presence of a uterus and at least one ovary.
* Ability and willingness to comply with study protocol.
* Have given written informed consent, prior to any study-related procedure, not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Inclusion Criteria for controls:

* Healthy females who have never been treated for cancer.
* Age between 11-35 and 40-50 years.
* Post-menarchal with regular cyclic menses (every 21-35 days)
* Presence of a uterus and at least 1 ovary.
* Ability and willingness to comply with study protocol.
* Have given written informed concent, prior to any study-related procedure, not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion Criteria:

* Current pregnancy.
* Use of hormonal contraception or use of hormone replacement therapy within the previous 4 weeks.
* Lactation within the previous 3 months.
* Chronic illness that would limit ability of participant to comply with study protocol.
* Any known medical condition, other than cancer, which in the judgement of the investigator is known to be associated with premature ovarian failure (such as Turner's Syndrome or Fragile X) or ovulatory dysfunction (such as thyroid disease, adrenal dysfunction, Cushing's syndrome, hyperprolactinemia, and polycystic ovarian syndrome).
* For controls, a history of infertility.

Ages: 11 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects with a history of cancer, or other conditions treated by chemotherapy, will be identified through local survivorship programs or self-referral. In addition, two groups of regularly menstruating unexposed subjects will be recruited through local advertising: a group of similar-age subjects and another group in the late reproductive years. Exposed and unexposed controls will be frequency matched with respect to age (within 2 years) at enrollment. In addition,subjects will be balanced with respect to self reported race/ethnicity. Enrollment is purposefully targeted and stratified for this study to reflect the population in the pediatric and adult oncology practices.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Reproductive hormones | Annually for 3-5 years
  Primary Outcomes for this study will include mean and changes in reproductive hormone measures obtained during the early follicular phase of the menstrual cycle (days 1-4).

SECONDARY OUTCOMES:
Antral Follicle Counts | Annually for 3-5 years
  All ovarian follicles and cysts will be measured by transvaginal or transabdominal ultrasound. Follicles will be measured in millimeters and grouped according to size: 2-5 mm, 6-9 mm, and >10 mm in diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa R Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Penn Reproductive Research Unit, 3701 Market Street, Suite 810, Philadelphia, Pennsylvania
  - Penn Medicine at Radnor, 250 King of Prussia Road, Radnor, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data will be shared with Dr. Jill Ginsberg, a co-investigator of the study.

REFERENCES:
- [Background] Gracia CR, Sammel MD, Freeman E, Prewitt M, Carlson C, Ray A, Vance A, Ginsberg JP. Impact of cancer therapies on ovarian reserve. Fertil Steril. 2012 Jan;97(1):134-40.e1. doi: 10.1016/j.fertnstert.2011.10.040. Epub 2011 Dec 2. PMID 22137491
- See also: Select "Clinical Trials" for Current Studies at Penn's Women's Health Clinical Research Center.For more information about participating in one of Penn Fertility Care's research studies please call 1-800-789-PENN. — http://www.pennmedicine.org/fertility/